CLINICAL TRIAL: NCT00822172
Title: Evaluation of Cilostazol in Combination With L-Carnitine in Subjects With Intermittent Claudication
Brief Title: Evaluation of Cilostazol in Combination With L-Carnitine
Acronym: ECLECTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CPC-08-01
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication; Peripheral Arterial Disease
Keywords: Peripheral Vascular Disease; Peripheral Arterial Disease; Intermittent Claudication; Peak Walking Time; Claudication Onset Time; Cilostazol; Carnitine
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Peripheral Arterial Disease | interventions — Carnitine; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol + L-Carnitine (Active Comparator): 1 tablet cilostazol 100 mg PO BID and 3 capsules L-carnitine 334 mg PO BID
  Interventions: Dietary Supplement: Levocarnitine tartrate; Drug: cilostazol
- Cilostazol + Placebo (Placebo Comparator): 1 tablet cilostazol 100 mg PO BID and 3 capsules placebo PO BID
  Interventions: Drug: cilostazol

INTERVENTIONS:
Dietary Supplement: Levocarnitine tartrate — Capsule form, 1,002 mg (3 capsules) taken by mouth two times per day (morning and evening). L-carnitine will be taken from Day 0 to Day 180.
  Other Names: Carnitine; L-carnitine; Levocarnitine
  Arms: Cilostazol + L-Carnitine
Drug: cilostazol — Background therapy beginning at 50mg (1 pill) taken by mouth two times per day for two to three weeks. Then 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for one to two weeks.
  Randomized therapy will consist of 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for approximately 180 days.
  Other Names: Pletal

SUMMARY:
The purpose of this study is to see how safe and effective L carnitine taken with cilostazol is compared to placebo taken with cilostazol for people with intermittent claudication. A second purpose of the study is to see if L-carnitine is absorbed into the blood stream.

DETAILED DESCRIPTION:
Peripheral Artery Disease (PAD) is a narrowing of the blood vessels that supply the leg with blood. It is caused by atherosclerosis (hardening of the arteries).

Muscles require oxygen carried by the blood. When the leg muscles do not get enough blood and oxygen, this can cause pain, cramping, fatigue, and/or discomfort in the leg muscles during walking or exercise. These symptoms are called intermittent claudication (IC). In more severe cases, tissues do not get enough blood and oxygen at rest, and pain may also be present when the legs are resting. Peripheral Artery Disease (PAD)is one of the most common causes of pain and disability in people between 55 and 75 years of age.

Cilostazol is a medication currently available by prescription for intermittent claudication. L-carnitine is an over-the-counter supplement. It is a natural substance in the human body and is also in some red meats, nuts, and energy drinks.

Some subjects in the study will take L-carnitine with cilostazol and others will take placebo with cilostazol. The purpose of this study is to see how safe and effective L carnitine taken with cilostazol is compared to placebo taken with cilostazol for people with intermittent claudication. A placebo is a tablet or pill that looks like regular medication, but it doesn't have any actual medicine in it. A second purpose of the study is to see if L-carnitine is absorbed into the blood stream.

ELIGIBILITY:
Inclusion Criteria:

* The subject is >40 years old.
* The subject has a diagnosis of Intermittent Claudication (IC) due to Peripheral Artery Disease (PAD).
* Ankle brachial index (ABI) < 0.90 in at least one extremity, or if Ankle brachial index (ABI)is ≥ 0.90 to ≤ 1.0, a reduction of at least 20% in Ankle brachial index (ABI), in at least one extremity, when measured within 1 minute after claudication-limiting treadmill testing. If the subject has non-compressible arteries then a toe brachial index (TBI) < 0.70 is required in at least one extremity.
* Symptoms of Intermittent Claudication (IC)must be stable for at least 3 months prior to Screening 1.
* Peak Walking Time (PWT) of ≥ 1 to ≤ 12 minutes on a Gardner protocol at Screening 2.
* If the subject is currently on statin therapy, they need to have been on statin therapy for at least 3 months prior to Screening 1. Subjects who have recently discontinued statin therapy must "wash-out" for at least one month prior to Screening 1.
* Tolerance to background therapy of cilostazol (approximately 2 weeks of 50 mg by mouth (PO) twice daily (BID), approximately 1 week of 100 mg PO BID) between Screening 2 and Baseline Visit.
* Subjects must be either male or females that are post-menopausal, surgically incapable of bearing children or if they are of childbearing potential must have a negative serum pregnancy test at Screening 1 and a negative urine pregnancy test at Day 0 and must agree to use double-barrier contraceptive methods until the end of investigational therapy (Day 180 Visit).
* The subject is able to comply with scheduled visits, treatment plan and laboratory tests.
* The subject is willing to participate in this study as documented by written informed consent.
* During the tolerance phase of the Screening period, the subject demonstrates at least 70% compliance with cilostazol and is willing to continue treatment.

Exclusion Criteria:

* Evidence of critical limb ischemia (CLI) (e.g., ischemic rest pain or ischemic ulceration).
* The subject has had a major amputation of the leg or any other amputation that limits walking ability.
* The subject has diabetes mellitus type 1 or poorly controlled diabetes mellitus type 2 (hemoglobin A1c (HbA1c) > 10).
* The subject has had a transient ischemic attack (TIA) or deep vein thrombosis in the last 3 months.
* The subject has had a stroke within the last 6 months.
* The subject has participated in an angiogenic gene therapy study, unless known to be given placebo.
* The subject has any of the following laboratory parameters at Screening 1:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin >3 times the upper limit of normal (ULN)
  * Serum creatinine >2.5 mg/dL
  * Hemoglobin (Hb) <10 g/dL
  * White blood cell (WBC) count <3.0 x 103/µL; or > 15 x 103/µL
  * Platelet count <100 x 103/µL
* The subject walks less than 1 minute at 2 miles per hour (mph), 0% grade as determined during the Screening 1 treadmill familiarization.
* The subject has clinically significant electrocardiogram (ECG) abnormalities at rest or changes during exercise or post-exercise at Screening 2 or Day 0.
* The subject has any history or clinical evidence of congestive heart failure (CHF), with which the clinician-investigator concurs.
* The subject has uncontrolled hypertension (resting blood pressure (BP) > 180/100 mmHg) or uncontrolled arrhythmic disorders at Screening 1.
* History of coronary or peripheral revascularization within 6 months prior to Screening 1.
* The subject plans to undergo coronary or peripheral revascularization during the course of the study.
* The subject is currently taking L-carnitine or medication for claudication (including pentoxifylline or cilostazol). In this situation, the subject would become eligible for Screening 1 after a 6 week washout of the medication.
* Subjects currently taking or those who anticipate taking ketoconazole, itraconazole, or erythromycin. The subject would become eligible for Screening 1 immediately after completion of therapy or discontinuation of the drug(s).
* The subject has a known, active malignancy that requires active anti-neoplastic therapy. (stable basal cell skin cancer allowed. Cancer being treated soley with hormonal therapy is allowed.)
* The subject has a severe co-morbidity with an expected survival of less than 2 years.
* The subject's Peak Walking Time (PWT) is limited by symptoms other than claudication (e.g., shortness of breath (SOB), fatigue, angina, arthritis, etc.). If, in the opinion of the investigator, the subject were to improve their Peak Walking Time (PWT) from study therapy to the extent that his or her walking would then be limited by a symptom other than claudication, the subject should not be enrolled.
* The subject has a history of alcohol or other substance abuse within 6 months of Screening 1.
* The subject has an inability to tolerate oral medication administration.
* The subject has a known or suspected allergy to the study medication(s) or class of study medication(s) (cilostazol or L-carnitine) to be administered.
* The subject has initiated an exercise training program within 3 months of Screening 1, has the inability to maintain his or her current level of physical activity throughout the study, or the subject plans on enrolling in an exercise training program during the study.
* The subject plans to change his/her smoking status during the planned duration of this study (subjects will be advised that stopping smoking is best for his/her health).
* The subject is currently pregnant or breastfeeding.
* The subject has received an investigational drug or biological agent within 30 days prior to Screening 1.
* The subject is currently participating in or plans to enroll in another clinical trial during this study.
* The subject has any other clinically significant medical or psychiatric condition that in the opinion of the Investigator could impact the subject's ability to successfully complete this trial.
* In the Investigator's opinion, the subject experienced any Adverse Events (AEs) during the tolerance phase of the Screening period that present a potential ongoing safety concern.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Goldenberg, MD, PhD, Study Chair — University of Colorado Heather Sciences Center
Locations (24):
- United States (24):
  - Internal Medicine Physicians Associates, Phoenix, Arizona
  - Tatum Ridge Internal Medicine, Phoenix, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California at Davis Vascular Center, Sacramento, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - Apex Research Institute, Santa Ana, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - DMI Healthcare Group, Inc., Pinellas Park, Florida
  - Meridian Research, St. Petersburg, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - HPV Heart, PA, Columbia, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester Medical Center, Rochester, New York
  - Durham VA-Medical Center, Durham, North Carolina
  - Radiant Research, Inc, Columbus, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Peripheral Vascular Associates, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research- Salt Lake City, Salt Lake City, Utah
  - Beloit Clinic Research Office, Beloit, Wisconsin

REFERENCES:
- [Background] Hiatt WR. Carnitine and peripheral arterial disease. Ann N Y Acad Sci. 2004 Nov;1033:92-8. doi: 10.1196/annals.1320.008. PMID 15591006
- [Background] Hiatt WR, Nawaz D, Brass EP. Carnitine metabolism during exercise in patients with peripheral vascular disease. J Appl Physiol (1985). 1987 Jun;62(6):2383-7. doi: 10.1152/jappl.1987.62.6.2383. PMID 3610932
- [Background] Hiatt WR. Management of Intermittent Claudication. Contemporary Diagnosis and management of Peripheral arterial Disease. 1 ed. Newtown: Handvbooks in Healthcare Co., Inc., 2004:51-9
- [Background] Rowlands TE, Donnelly R. Medical therapy for intermittent claudication. Eur J Vasc Endovasc Surg. 2007 Sep;34(3):314-21. doi: 10.1016/j.ejvs.2007.04.001. Epub 2007 May 29. PMID 17532651
- [Background] Dawson DL, Cutler BS, Meissner MH, Strandness DE Jr. Cilostazol has beneficial effects in treatment of intermittent claudication: results from a multicenter, randomized, prospective, double-blind trial. Circulation. 1998 Aug 18;98(7):678-86. doi: 10.1161/01.cir.98.7.678. PMID 9715861
- [Background] Money SR, Herd JA, Isaacsohn JL, Davidson M, Cutler B, Heckman J, Forbes WP. Effect of cilostazol on walking distances in patients with intermittent claudication caused by peripheral vascular disease. J Vasc Surg. 1998 Feb;27(2):267-74; discussion 274-5. doi: 10.1016/s0741-5214(98)70357-x. PMID 9510281
- [Background] Elam MB, Heckman J, Crouse JR, Hunninghake DB, Herd JA, Davidson M, Gordon IL, Bortey EB, Forbes WP. Effect of the novel antiplatelet agent cilostazol on plasma lipoproteins in patients with intermittent claudication. Arterioscler Thromb Vasc Biol. 1998 Dec;18(12):1942-7. doi: 10.1161/01.atv.18.12.1942. PMID 9848888
- [Background] Beebe HG, Dawson DL, Cutler BS, Herd JA, Strandness DE Jr, Bortey EB, Forbes WP. A new pharmacological treatment for intermittent claudication: results of a randomized, multicenter trial. Arch Intern Med. 1999 Sep 27;159(17):2041-50. doi: 10.1001/archinte.159.17.2041. PMID 10510990
- [Background] Dawson DL, Cutler BS, Hiatt WR, Hobson RW 2nd, Martin JD, Bortey EB, Forbes WP, Strandness DE Jr. A comparison of cilostazol and pentoxifylline for treating intermittent claudication. Am J Med. 2000 Nov;109(7):523-30. doi: 10.1016/s0002-9343(00)00569-6. PMID 11063952
- [Background] Strandness DE Jr, Dalman RL, Panian S, Rendell MS, Comp PC, Zhang P, Forbes WP. Effect of cilostazol in patients with intermittent claudication: a randomized, double-blind, placebo-controlled study. Vasc Endovascular Surg. 2002 Mar-Apr;36(2):83-91. doi: 10.1177/153857440203600202. PMID 11951094
- [Background] Regensteiner JG, Ware JE Jr, McCarthy WJ, Zhang P, Forbes WP, Heckman J, Hiatt WR. Effect of cilostazol on treadmill walking, community-based walking ability, and health-related quality of life in patients with intermittent claudication due to peripheral arterial disease: meta-analysis of six randomized controlled trials. J Am Geriatr Soc. 2002 Dec;50(12):1939-46. doi: 10.1046/j.1532-5415.2002.50604.x. PMID 12473004
- [Background] Thompson PD, Zimet R, Forbes WP, Zhang P. Meta-analysis of results from eight randomized, placebo-controlled trials on the effect of cilostazol on patients with intermittent claudication. Am J Cardiol. 2002 Dec 15;90(12):1314-9. doi: 10.1016/s0002-9149(02)02869-2. PMID 12480040
- [Background] Pratt CM. Analysis of the cilostazol safety database. Am J Cardiol. 2001 Jun 28;87(12A):28D-33D. doi: 10.1016/s0002-9149(01)01719-2. PMID 11434897
- [Background] Hiatt WR, Money SR, Brass EP. Long-term safety of cilostazol in patients with peripheral artery disease: the CASTLE study (Cilostazol: A Study in Long-term Effects). J Vasc Surg. 2008 Feb;47(2):330-336. doi: 10.1016/j.jvs.2007.10.009. Epub 2007 Dec 26. PMID 18155871
- [Background] Hiatt WR, Regensteiner JG, Creager MA, Hirsch AT, Cooke JP, Olin JW, Gorbunov GN, Isner J, Lukjanov YV, Tsitsiashvili MS, Zabelskaya TF, Amato A. Propionyl-L-carnitine improves exercise performance and functional status in patients with claudication. Am J Med. 2001 Jun 1;110(8):616-22. doi: 10.1016/s0002-9343(01)00704-5. PMID 11382369
- [Background] Muller DM, Seim H, Kiess W, Loster H, Richter T. Effects of oral L-carnitine supplementation on in vivo long-chain fatty acid oxidation in healthy adults. Metabolism. 2002 Nov;51(11):1389-91. doi: 10.1053/meta.2002.35181. PMID 12404185
- [Background] Brass EP, Anthony R, Cobb FR, Koda I, Jiao J, Hiatt WR. The novel phosphodiesterase inhibitor NM-702 improves claudication-limited exercise performance in patients with peripheral arterial disease. J Am Coll Cardiol. 2006 Dec 19;48(12):2539-45. doi: 10.1016/j.jacc.2006.07.064. Epub 2006 Nov 28. PMID 17174195
- [Background] Hiatt WR, Hirsch AT, Regensteiner JG, Brass EP. Clinical trials for claudication. Assessment of exercise performance, functional status, and clinical end points. Vascular Clinical Trialists. Circulation. 1995 Aug 1;92(3):614-21. doi: 10.1161/01.cir.92.3.614. No abstract available. PMID 7634476
- [Background] Rizza v, Lorefice R, Rizza N et al. Pharmacokinetics of L-Carnitine in Human Subjects. In: Ferrari R, DiMauro S, Sherwood G, eds. L-Carnitine and its Role in Medicine: From Function to Therapy. 1 ed San Diego: Academic Press, Inc., 1992:63-77.
- [Background] Hiatt WR, Wolfel EE, Regensteiner JG, Brass EP. Skeletal muscle carnitine metabolism in patients with unilateral peripheral arterial disease. J Appl Physiol (1985). 1992 Jul;73(1):346-53. doi: 10.1152/jappl.1992.73.1.346. PMID 1506390
- [Background] Brevetti G, Angelini C, Rosa M, Carrozzo R, Perna S, Corsi M, Matarazzo A, Marcialis A. Muscle carnitine deficiency in patients with severe peripheral vascular disease. Circulation. 1991 Oct;84(4):1490-5. doi: 10.1161/01.cir.84.4.1490. PMID 1914091
- [Background] Bauer TA, Brass EP, Hiatt WR. Impaired muscle oxygen use at onset of exercise in peripheral arterial disease. J Vasc Surg. 2004 Sep;40(3):488-93. doi: 10.1016/j.jvs.2004.06.025. PMID 15337878
- [Background] Bauer TA, Brass EP, Barstow TJ, Hiatt WR. Skeletal muscle StO2 kinetics are slowed during low work rate calf exercise in peripheral arterial disease. Eur J Appl Physiol. 2007 May;100(2):143-51. doi: 10.1007/s00421-007-0412-0. Epub 2007 Feb 20. PMID 17310391
- [Background] Brass EP, Hiatt WR, Gardner AW, Hoppel CL. Decreased NADH dehydrogenase and ubiquinol-cytochrome c oxidoreductase in peripheral arterial disease. Am J Physiol Heart Circ Physiol. 2001 Feb;280(2):H603-9. doi: 10.1152/ajpheart.2001.280.2.H603. PMID 11158957
- [Background] Brass EP. Supplemental carnitine and exercise. Am J Clin Nutr. 2000 Aug;72(2 Suppl):618S-23S. doi: 10.1093/ajcn/72.2.618S. PMID 10919968
- [Background] Hiatt WR, Regensteiner JG, Wolfel EE, Ruff L, Brass EP. Carnitine and acylcarnitine metabolism during exercise in humans. Dependence on skeletal muscle metabolic state. J Clin Invest. 1989 Oct;84(4):1167-73. doi: 10.1172/JCI114281. PMID 2794054
- [Background] Eder K, Felgner J, Becker K, Kluge H. Free and total carnitine concentrations in pig plasma after oral ingestion of various L-carnitine compounds. Int J Vitam Nutr Res. 2005 Jan;75(1):3-9. doi: 10.1024/0300-9831.75.1.3. PMID 15830915
- [Background] Rubin MR, Volek JS, Gomez AL, Ratamess NA, French DN, Sharman MJ, Kraemer WJ. Safety measures of L-carnitine L-tartrate supplementation in healthy men. J Strength Cond Res. 2001 Nov;15(4):486-90. PMID 11726261
- [Background] Giamberardino MA, Dragani L, Valente R, Di Lisa F, Saggini R, Vecchiet L. Effects of prolonged L-carnitine administration on delayed muscle pain and CK release after eccentric effort. Int J Sports Med. 1996 Jul;17(5):320-4. doi: 10.1055/s-2007-972854. PMID 8858401
- [Background] Volek JS, Kraemer WJ, Rubin MR, Gomez AL, Ratamess NA, Gaynor P. L-Carnitine L-tartrate supplementation favorably affects markers of recovery from exercise stress. Am J Physiol Endocrinol Metab. 2002 Feb;282(2):E474-82. doi: 10.1152/ajpendo.00277.2001. PMID 11788381
- [Background] Kraemer WJ, Volek JS, French DN, Rubin MR, Sharman MJ, Gomez AL, Ratamess NA, Newton RU, Jemiolo B, Craig BW, Hakkinen K. The effects of L-carnitine L-tartrate supplementation on hormonal responses to resistance exercise and recovery. J Strength Cond Res. 2003 Aug;17(3):455-62. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 12930169
- [Background] Spiering BA, Kraemer WJ, Vingren JL, Hatfield DL, Fragala MS, Ho JY, Maresh CM, Anderson JM, Volek JS. Responses of criterion variables to different supplemental doses of L-carnitine L-tartrate. J Strength Cond Res. 2007 Feb;21(1):259-64. doi: 10.1519/00124278-200702000-00046. PMID 17313301
- [Background] Brevetti G, Chiariello M, Ferulano G, Policicchio A, Nevola E, Rossini A, Attisano T, Ambrosio G, Siliprandi N, Angelini C. Increases in walking distance in patients with peripheral vascular disease treated with L-carnitine: a double-blind, cross-over study. Circulation. 1988 Apr;77(4):767-73. doi: 10.1161/01.cir.77.4.767. PMID 3280157
- [Background] Brevetti G, Perna S, Sabba C, Rossini A, Scotto di Uccio V, Berardi E, Godi L. Superiority of L-propionylcarnitine vs L-carnitine in improving walking capacity in patients with peripheral vascular disease: an acute, intravenous, double-blind, cross-over study. Eur Heart J. 1992 Feb;13(2):251-5. doi: 10.1093/oxfordjournals.eurheartj.a060155. PMID 1555624
- [Background] Brevetti G, Diehm C, Lambert D. European multicenter study on propionyl-L-carnitine in intermittent claudication. J Am Coll Cardiol. 1999 Nov 1;34(5):1618-24. doi: 10.1016/s0735-1097(99)00373-3. PMID 10551714
- [Derived] Goldenberg NA, Krantz MJ, Hiatt WR. L-Carnitine plus cilostazol versus cilostazol alone for the treatment of claudication in patients with peripheral artery disease: a multicenter, randomized, double-blind, placebo-controlled trial. Vasc Med. 2012 Jun;17(3):145-54. doi: 10.1177/1358863X12442264. PMID 22615190
- See also: CPC Home Page — http://www.cpcmed.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was randomized on September 19th, 2008 and the last subject was randomized on May 7, 2010. Clinical study sites were a mixture of university/hospital settings, Veteran Affairs hospitals, professional research centers and medical clinics.
Pre-assignment Details: The study included a cilostazol run in period. From the 164 participants who remained eligible at the end of the run in period, only 1 participant did not subsequently receive treatment. This was due to voluntary withdrawal by the participant.
Groups:
- Cilostazol + L-Carnitine: Levocarnitine tartrate : Capsule form, 1,002 mg (3 capsules) taken by mouth two times per day (morning and evening). L-carnitine will be taken from Day 0 to Day 180.
  cilostazol : Background therapy beginning at 50mg (1 pill) taken by mouth two times per day for two to three weeks. Then 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for one to two weeks.
  Randomized therapy will consist of 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for approximately 180 days.
- Cilostazol + Placebo: cilostazol : Background therapy beginning at 50mg (1 pill) taken by mouth two times per day for two to three weeks. Then 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for one to two weeks.
  Randomized therapy will consist of 100 mg (1 pill) to be taken by mouth two times per day (morning and evening) for approximately 180 days.
Period: Overall Study
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Started | 80 | 83
Completed | 65 | 64
Not Completed | 15 | 19
Not completed — Adverse Event | 10 | 12
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — site closed | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo | Total
Number analyzed (Participants) | 80 | 83 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 27 | 70
  >=65 years | 37 | 56 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.39) | 67.3 (8.00) | 66.5 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 66 | 67 | 133
Region of Enrollment [Number; unit: participants]
  United States | 80 | 83 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Walking Time (PWT) at Day 180
Description: Subjects were asked to complete a standardized exercise treadmill test using a modified Gardner protocol. Subjects walked on the treadmill until they were physically unable to walk further either as a result of their peripheral artery disease (PAD) symptoms or other non-PAD symptoms. This maximum time walked is referred to as the peak walking time (PWT) and reported in minutes/seconds. The exercise treadmill test was conducted at Screening, Baseline, Day 90, and Day 180 visits. The log transformation is used to make highly skewed distributions less skewed.
Time Frame: Baseline, Day 180
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: Log Minutes
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 74 | 71
Log Minutes | 0.241 (0.3836) | 0.134 (0.3343)
Statistical Analysis 1: Comparison: Cilostazol + L-Carnitine vs Cilostazol + Placebo; Test type: Superiority; p = 0.076, two-sample equal-variances t-test

2. Secondary Outcome: Change From Baseline in Peak Walking Time at Day 180
Description: as for outcome 1
Time Frame: Baseline, Day 180
Population: Per Protocol (PP) Population
Measure: Mean (Standard Deviation); unit: Log Minutes
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 60 | 58
Log Minutes | 0.267 (0.3516) | 0.145 (0.3124)
Statistical Analysis 1: Comparison: Cilostazol + L-Carnitine vs Cilostazol + Placebo; Test type: Superiority; p = 0.048, two-sample equal-variances t-test

3. Secondary Outcome: Change From Baseline in Peak Walking Time at Day 90
Description: as for outcome 1
Time Frame: Baseline, Day 90
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: Log Minutes
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 69 | 65
Log Minutes | 0.166 (0.3571) | 0.139 (0.3293)
Statistical Analysis 1: Comparison: Cilostazol + L-Carnitine vs Cilostazol + Placebo; Test type: Superiority; p = 0.650, two-sample equal-variances t-test

4. Secondary Outcome: Change From Baseline in Claudication Onset Time at Day 180
Description: Subjects were asked to complete a standardized exercise treadmill test using a modified Gardner protocol. Subjects walked on the treadmill until they were physically unable to walk further either as a result of their peripheral artery disease (PAD) symptoms or other non-PAD symptoms. The time during the conduct of the exercise treadmill test at which the subject first reported claudication symptoms is referred to as the claudication onset time (COT) and reported in minutes/seconds. The exercise treadmill test was conducted at Screening, Baseline, Day 90, and Day 180 visits. The log transformation is used to make highly skewed distributions less skewed.
Time Frame: Baseline, Day 180
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: Log Minutes
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 66 | 66
Log Minutes | 1.065 (0.6680) | 0.896 (0.7364)

5. Secondary Outcome: Change From Baseline in Claudication Onset Time at Day 90
Description: as for outcome 4
Time Frame: Baseline, Day 90
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: Log Minutes
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 68 | 63
Log Minutes | 1.001 (0.6476) | 0.815 (0.7000)

6. Secondary Outcome: Change From Baseline in Walking Impairment Questionnaire for Walking Distance at Day 180
Description: Subjects completed the Walking Impairment Questionnaire (WIQ) whereby they were asked about their maximal walking distance before having to rest as a result of claudication symptoms associated with their peripheral artery disease (PAD). The WIQ was administered at the Baseline, Day 90, and Day 180 visits. On the WIQ subjects were asked a series of questions related to their degree of physical difficulty that best described how hard it was for the subject to walk on level ground without stopping to rest. The questions began by asking the degree of difficulty walking around indoors, then 50 feet, 150 feet, 300 feet, 600 feet, 900 feet, and lastly 1500 feet. The responses range from None (best outcome) to Slight, then Some, then Much, then lastly Unable (worst outcome). The walking distance score was calculated from the 7 questions in the section by way of a weighted sum. A score of 100 indicated no walking impairment. A score of 0 corresponded to the highest degree of walking impairment
Time Frame: Baseline, Day 180
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 68 | 68
score on a scale | 13.20 (22.001) | 6.57 (24.288)

7. Secondary Outcome: Change From Baseline in Walking Impairment Questionnaire for Walking Distance at Day 90
Description: as for outcome 6
Time Frame: Baseline, Day 90
Population: modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Number analyzed (Participants) | 71 | 66
score on a scale | 12.98 (25.251) | 10.01 (21.354)

ADVERSE EVENTS:
Arm/Group | Cilostazol + L-Carnitine | Cilostazol + Placebo
Serious Adverse Events (participants affected / at risk) | 11/80 | 10/83
Other Adverse Events (participants affected / at risk) | 19/80 | 22/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol + L-Carnitine (N=80) | Cilostazol + Placebo (N=83)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Prostate cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
Urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (General disorders) | 2 (2) | 0 (0)
Ureteric fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Endocrine disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol + L-Carnitine (N=80) | Cilostazol + Placebo (N=83)
Diarrhoea (Gastrointestinal disorders) | 9 (16) | 8 (17)
Headache (Nervous system disorders) | 10 (15) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes